CLINICAL TRIAL: NCT00707720
Title: Multi-center Feasibility Study to Evaluate the Safety of the Trans-oral Endoscopic Restrictive Implant System (TERIS) for the Treatment of Obesity
Brief Title: Multi-Center Feasibility Study of Trans-oral Endoscopic Restrictive Implant System (TERIS) for Treatment of Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BaroSense Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSI 07-01
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TERIS procedure (Experimental): TERIS procedure for the treatment of obesity
  Interventions: Device: TERIS procedure

INTERVENTIONS:
Device: TERIS procedure — The implantation of the restrictive implant

SUMMARY:
The Barosense Trans-oral Endoscopic Restrictive Implant System (TERIS) is an investigational system being evaluated for safety The system uses endoscopic guidance to trans-orally implant a restrictive reservoir for food entering the stomach in obese and morbidly obese subjects to induce early and prolonged satiety. The Intended Use of the system is for the treatment of obesity.

DETAILED DESCRIPTION:
Obesity is now considered to be epidemic through most of the industrialized world. The consequences of obesity on long-term health of individuals is now well documented. While lifestyle changes in diet and activity level are the key instruments to arresting or reversing this condition, conventional medically supervised programs have proven only marginally effective. Bariatric surgery has shown to be a reliable long-term treatment for reducing excess body weight. Though surgical techniques have evolved and complication rates have been reduced, surgery on these patients still carries significant mortality and morbidity.

Techniques and instruments are now being developed to allow for Endoscopic approaches to these procedures that will aim to reduce the complications associated with open or laparoscopic technique for these procedures.

The primary objective of this study is to evaluate the safety of the Trans-oral Endoscopic Restrictive Implant System (TERIS) procedure for the treatment of obesity over a six month follow-up period.

A secondary objective is to perform a preliminary evaluation of the efficacy of the TERIS procedure in order to guide the design of future studies, including a pivotal trial.

This is a prospective feasibility study at up to 3 investigational sites of up to 40 subjects who are obese and have failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone, or in combination. Up to 60 subjects may be enrolled, and undergo baseline evaluation in order to obtain a final total of up to 40 subjects appropriate for trans-oral implant. Barosense intends to use data from this study in support of subsequent investigational studies, including a pivotal trial

ELIGIBILITY:
Inclusion Criteria:

* All of the following criteria must be met for study participation/device implantation:

  1. Subject, male or female, is age 18 to 50 years of age.
  2. Subject must be able to understand and be willing to sign an informed consent document.
  3. Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
  4. Subject has a BMI of 40.0-49.0 or has a BMI of 35.0-39.9 plus one or more co-morbid diseases expected to improve with weight loss (e.g. hypertension, dyslipidemia, obstructive sleep apnea, or diabetes mellitus).
  5. Subject must be fully ambulatory, without chronic reliance on walking aids such as crutches, walkers or a wheelchair.
  6. Subject must be of sufficient and stable medical health, as evaluated by the Principal Investigator.
  7. Subject must have a primary care physician that will manage the subject for any co-morbid conditions throughout the study.
  8. Subject must have failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination.
  9. Subject agrees to refrain from any type of reconstructive surgery that may affect body weight such as mammoplasty or abdominal lipoplasty or liposuction, during the trial.

Exclusion Criteria:

A subject is ineligible to participate in this study if they meet any of the following criteria:

1. Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease.
2. Subject has an A1C ≥ 7.0%, or other indicator of poorly controlled diabetes.
3. Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
4. Subject has pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
5. Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility.
6. Subject has renal and/or hepatic insufficiency.
7. Subject has thyroid disease which is not controlled with medication.
8. Subject has a history of intestinal strictures or adhesions.
9. Subject has systemic infection in the body at the time of TERIS procedure.
10. Female subject who is pregnant (i.e., has a positive urine or blood pregnancy test prior to device implant), is suspected to be pregnant, is lactating or is of childbearing potential but refuses to use adequate contraception during the study.
11. Subject has had previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy; gastrointestinal tumors; esophageal or gastric varices, or gastroparesis.
12. Subject has severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000) or is presently taking heparin, coumadin, warfarin, or other anticoagulants or other medications which impede coagulation or platelet aggregation.
13. Subjects who are unable to discontinue use of aspirin and/or non-steroidal anti-inflammatory agents (NSAIDs) at least 14 days prior to a device implant or device removal procedure and continuing for 14 days post-procedure(s).
14. Subjects undergoing chronic steroid therapy.
15. Subjects undergoing immunosuppressive therapy.
16. Subjects who cannot discontinue either prescription or over the counter weight loss medications for at least 30 days prior to the procedure as well as during the trial period.
17. Subjects who have cardiac pacemakers or other electronic implantable devices.
18. Subjects who have hiatal hernias greater than 2 cm.
19. Subjects who have poorly controlled psychiatric disease including but not limited to manic-depressive disorder, schizophrenia, borderline personality disorder, depression or suicidal tendencies.
20. Subject has Crohn's disease or Ulcerative Colitis.
21. Subject currently uses or has a history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
22. Subject has participated in a clinical study with an investigational new drug, biological, or therapeutic device within £ 28 days prior to enrollment in this study, and does not agree to abstain from participation in other clinical trials of any kind during this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events relating to the procedure and device | 6 months

SECONDARY OUTCOMES:
Weight loss, Excess weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Stecco, MD, Study Director — Medical Consultant
Locations (1):
- Hopital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Biertho L, Hould FS, Lebel S, Biron S. Transoral endoscopic restrictive implant system: a new endoscopic technique for the treatment of obesity. Surg Obes Relat Dis. 2010 Mar 4;6(2):203-5. doi: 10.1016/j.soard.2009.08.006. Epub 2009 Aug 28. No abstract available. PMID 19796996